CLINICAL TRIAL: NCT07301151
Title: Feasibility of Using a Conversational Agent for Promoting Smoking Cessation Treatment Utilization
Brief Title: PASCAL Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00026782; P50MD017342 (NIH)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation; Smoking (Tobacco) Addiction
Keywords: cigarette smoking; chatbot
MeSH Terms: conditions — Smoking Cessation; Smoking; Behavior, Addictive; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chatbot assisted smoking trigger management (Experimental)
  Interventions: Other: chatbot
- control group (Active Comparator)
  Interventions: Other: no chatbot

INTERVENTIONS:
Other: chatbot — a chatbot will alert during predicted high risk smoking times and suggest approaches to manage potential smoking triggers
  Arms: chatbot assisted smoking trigger management
Other: no chatbot — no chatbot is provided
  Arms: control group

SUMMARY:
The goal of this randomized study is to assess if a conversational agent (or chatbot) that the investigators have developed to help with quitting smoking is acceptable to people trying to quit smoking and to also collect initial information regarding its effectiveness.

In this study, some participants trying to quit smoking will be provided with this chatbot while other participants will not be

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black or African American
* Be at least 21 years of age
* Meet a minimum smoking amount
* Be willing to make a quit attempt in the next 30 days
* Have a smartphone capable of downloading and running the study app
* Be able to upload data from the app
* Agree to receive text message reminders about study activities
* Be a native English speaker
* Reside in Minnesota.

Exclusion Criteria:

* Medicinal nicotine use would require careful monitoring by a healthcare professional
* Medical condition or medication used likely to significantly interfere with study outcomes or to be significantly affected by changes in smoking behavior
* Are pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of trial procedures | 1 day
  The proportion of enrolled participants who download the study app
Feasibility of study procedures | 2 weeks
  The proportion of participants (among those who downloaded the app) who complete the week 2 post-quit visit
Health Information Technology Usability Evaluation Scale (Health-ITUES) | 2 weeks
  This scale will be used to access the acceptability of study app. The scale consists of 20 questions scored from 1 to 5 with higher values indicating more positive response

SECONDARY OUTCOMES:
Average number of daily interactions with the study app | 2 weeks
The average number of cigarettes smoked per day | 2 weeks
Average number of nicotine lozenges used | 2 weeks
The proportion of participants who complete the week 8 post-quit visit | 8 weeks
The proportion of participants not smoking for the 7 day period before the week 2 visit | 2 weeks
The proportion of participants not smoking for the 7 day period before the week 8 visits | 8 weeks
The proportion of participants not smoking at all between the quit date and the week 2 visit | 2 weeks
The proportion of participants not smoking at all between the quit date and the week 8 visit | 8 weeks
Motivation to quit smoking | 2 weeks
  Using a 1 - 10 scale on the contemplation to quit ladder (1 - no interest in quitting; 10 - will never smoke again)
Brief Questionnaire of Smoking Urges (QSU-Brief) | 2 weeks
  Questionnaire assessing craving severity. Range for total score is 10 - 70 with higher score indicating greater craving
The Minnesota Nicotine Withdrawal Scale (MNWS) | 2 weeks
  Questionnaire assessing withdrawal symptom severity. Range for total score is 0 - 36 with higher score indicating greater withdrawal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data will be deposited into the University of Minnesota Data Repository (DRUM)